CLINICAL TRIAL: NCT05201222
Title: Predictive Value of Induced Sleep Endoscopy on Surgical Indication in Obstructive Sleep Apnea Syndromes
Acronym: SOMMEIL_INDUIT
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Institut Arthur Vernes (Unknown)
Responsible Party: Sponsor
Other Study IDs: SOMMEIL_INDUIT
Record Dates: First submitted 2021-12-31; First posted 2022-01-21 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obstructive sleep apnea syndrome (OSA) is a pathology that affects 2 to 15% of the French adult population and more than 30% of subjects over 65 years old. It consists of repeated collapses of the upper airways during sleep leading to interruptions in ventilation (apneas) or significant reductions in ventilation (hypopneas). Balagny et al. have demonstrated the occurrence of hypertension in patients screened positive for sleep apnea syndrome in a French general population cohort. It is also established that sleep apnea increases the risk of cardiovascular disorders, such as metabolic syndrome (combining abdominal obesity and metabolic disorders), hypertension, heart rhythm disorders, especially at night, atherosclerosis (deposits of atheromatous plaques on the artery walls) or type 2 diabetes. These different complications increase the risk of cardiovascular accidents such as cardiac arrest, myocardial infarction, stroke, and expose to a risk of premature death (Inserm). The treatment of choice is night-time positive pressure ventilation, made possible by the use of a breathing apparatus (Continuous Positive Airway Pressure or CPAP). Alternatives to CPAP are the use of a nocturnal Mandibular Advancement Orthosis (MAO) which advances the jaw and allows a pharyngeal opening, and surgery in selected patients. The phenomenon at the origin of apneas is due to a relaxation of the muscles of the pharyngeal wall located at different heights. This obstruction is favored by anatomical particularities specific to each individual. The clinical examination can detect certain anomalies (enlarged tonsils, obstructive soft palate, prominent tongue base, abnormal epiglottis) and propose surgery to remove the obstruction.

Nevertheless, it remains difficult to affirm that the detected anomaly is really at the origin of the obstruction and surgical failures are frequent. Endoscopy under induced sleep has been developed for about 10 years in France. This examination, widely used in the world, remains confidential in France. It consists, in the operating room, in inducing a medicated sleep (specific drugs delivered by an anesthetist) and performing a pharyngolaryngeal fibroscopy. The ENT physician can then visualize "live" the site and origin of the obstruction during an apnea.

The main objective is to evaluate the interest of endoscopy under sleep before making a surgical indication in a patient presenting a sleep apnea syndrome. The secondary objective is to evaluate the reliability of sleep endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient with sleep apnea syndrome confirmed by polysomnographic or polygraphic recording The parameters of interest (Apnea Hypopnea Index, percentage of snoring and desaturation during the recording) are collected and in an identical way by its two examinations. They differ by the recording of other parameters.
* Patient for whom a sleep endoscopy is performed: clinical/recording discordance, failure or intolerance of the proposed treatment (OAM, PPC); surgical indication for OSA (tonsillectomy and/or velopasty)
* French speaking patient

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with sleep apnea syndrome confirmed by polysomnographic or polygraphic recording, for whom a sleep endoscopy is performed: clinical/recording discordance, failure or intolerance of the proposed treatment (OAM, PPC); surgical indication for OSA (tonsillectomy and/or velopasty) between 11/12/2012 and 05/10/2020.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Interest of sleep endoscopy before making a surgical indication in a patient with sleep apnea syndrome | Day 1
  This outcome corresponds to the number of patients for whom the surgical indication was maintained according to the data collected during the sleep endoscopy.

SECONDARY OUTCOMES:
Reliability of endoscopy under sleep | Day 1
  This outcome corresponds to the comparison of the number of patients for whom the treatment considered before the sleep endoscopy and the type of treatment were finally performed.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent YONA, MD, Principal Investigator — Institut Arthur Vernes
Locations (1):
- Institut Arthur Vernes, Paris, France

REFERENCES:
- [Background] Chong KB, De Vito A, Vicini C. Drug-Induced Sleep Endoscopy in Treatment Options Selection. Sleep Med Clin. 2019 Mar;14(1):33-40. doi: 10.1016/j.jsmc.2018.11.001. Epub 2018 Dec 3. PMID 30709531
- [Background] De Vito A, Carrasco Llatas M, Ravesloot MJ, Kotecha B, De Vries N, Hamans E, Maurer J, Bosi M, Blumen M, Heiser C, Herzog M, Montevecchi F, Corso RM, Braghiroli A, Gobbi R, Vroegop A, Vonk PE, Hohenhorst W, Piccin O, Sorrenti G, Vanderveken OM, Vicini C. European position paper on drug-induced sleep endoscopy: 2017 Update. Clin Otolaryngol. 2018 Dec;43(6):1541-1552. doi: 10.1111/coa.13213. Epub 2018 Sep 30. PMID 30133943
- [Background] Aljassim A, Pang KP, Rotenberg BW. Does Drug-Induced Sleep Endoscopy Improve Sleep Surgery Outcomes? Laryngoscope. 2020 Nov;130(11):2518-2519. doi: 10.1002/lary.28668. Epub 2020 Apr 18. No abstract available. PMID 32304328
- [Background] Kezirian EJ, Hohenhorst W, de Vries N. Drug-induced sleep endoscopy: the VOTE classification. Eur Arch Otorhinolaryngol. 2011 Aug;268(8):1233-1236. doi: 10.1007/s00405-011-1633-8. Epub 2011 May 26. PMID 21614467
- [Background] Kotecha B, De Vito A. Drug induced sleep endoscopy: its role in evaluation of the upper airway obstruction and patient selection for surgical and non-surgical treatment. J Thorac Dis. 2018 Jan;10(Suppl 1):S40-S47. doi: 10.21037/jtd.2017.10.32. PMID 29445527
- See also: Prévalence du syndrome d'apnée du sommeil et son association avec les évènements cardiovasculaires dans la population générale française — https://www.em-consulte.com/article/1343329/prevalence-du-syndrome-d-apnee-du-sommeil-et-son-a